CLINICAL TRIAL: NCT01887041
Title: Quality of Life After Bilioenteric Anastomosis in Comparison to Endoscopically Placed Stents in Patients With Unresectable Pancreatic Cancer and Jaundice
Brief Title: Quality of Life After Biliodigestive Anastomosis (BDA) or Stents to Treat Biliary Obstruction in Pancreas Cancer
Acronym: BYPAPA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruiting problems
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1 - mtachezy
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Local Tumor Spread; Advanced Cancer; Metastasized; Pancreatic Cancer Non-resectable; Jaundice
Keywords: Advanced, metastasising pancreatic head carcinoma; Jaundice; Biliodigestive anastomosis; Endoscopically inserted biliary tract drainage; Quality of Life
MeSH Terms: conditions — Neoplasm Metastasis; Jaundice | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stent (Active Comparator): Arm B, after randomisation the biliary tract stents shall remain. The patients in study arm B will also receive chemotherapy and gemcitabine, according to the recommended palliative therapy for a pancreas carcinoma.
  Interventions: Procedure: Stent
- Biliodigestive anastomosis (Active Comparator): Study arm A will, after randomisation, have a biliodigestive anastomosis inserted. After the healing of the wound (al least 14 days postoperative) the treatment using gemcitabine, according to the plan mentioned below.
  Gemcitabine shall be administered on days 1, 8 and 15 of each 4 week cycle. The cycle is defined as a weekly, over a period of 3 consecutive weeks, applied infusions, followed by 1 week pause. On the day of therapy a dosage of 1000 mg/ml body surface shall be administered, intravenous, over a period of 30 minutes.
  Interventions: Procedure: Biliodigestive anastomosis

INTERVENTIONS:
Procedure: Stent — Endoscopically inserted biliary tract drainage
  Arms: Stent
Procedure: Biliodigestive anastomosis — Biliodigestive anastomosis
  Arms: Biliodigestive anastomosis

SUMMARY:
To compare the quality of life (QoL) in patients receiving a bilioenteric anastomosis vs. endoscopical stenting for palliation of biliary obstruction due to locally unresectable or metastatic pancreatic cancer. In the past, endoscopy seems to have been favoured based on older studies, but with new chemotherapeutic regimens available, the likelihood to experience stent complications has increased. Therefore, the issue as to which palliation should be favoured has to be reconsidered.

DETAILED DESCRIPTION:
The aim of this multi-centre, prospective-randomised study was to compare the effectiveness of palliative applications on patients suffering from a local, advanced and/or hepatic, metastasising, non-resectable pancreas head carcinoma and jaundice.

Before randomisation, all patients are fitted with an endoscopically inserted biliary tract drainage endoscopically inserted. When postoperatively ascertained that the pancreas head carcinoma is non-resectable, the patient shall be electronically registered and randomly assigned to one of the palliative strategies. Group 1 will be fitted with a biliodigestive anastomosis. Group 2 will continue with the endoscopically inserted drainage. Regardless of which group they belong to, all patients will receive a palliative chemotherapy.

The primary parameter is the average quality of life over a period of 6 months post-operatively, to be analysed monthly using identical questionnaires. The comparison of the randomisation groups will be carried out using a co-variance analysis (ANCOVA) with the initial value, taken directly before the operation, to be used as co-variant.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient with local, advanced adenocarcinoma of the pancreas head and jaundice.
2. Performance-status of 50 or above on the Karnofsky-scale (see attachment).
3. Adequate bone marrow reserves: leukocyte level > 3.5 x 10´/l, thrombocyte level level > 100 x 10/l; Haemoglobin> 80g/l.
4. Male or female patients, at least 18 years old.
5. Women of child bearing age must be sufficient protected against pregnancy (contraception) during and for 3 months after the end of the study.

Exclusion Criteria:

1. Adult patients with focal, advanced adenocarcinoma of the pancreas head and no jaundice; also no jaundice in their anamnesis and with no endoscopic retrograde cholangio-pancreaticography (ERCP)-induced intervention.
2. Pregnancy
3. Breast feeding
4. Contra-indication for gemcitabine

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Outcome of Quality of Life. | 2 1/2 years

SECONDARY OUTCOMES:
The incidence of surgical complications and complications, with regard to the endo-scopic stent insertion, are further aspects that shall be examined in this study. | 2 1/2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jacob R Izbicki, MD, Principal Investigator — Universitätsklinik Hamburg
Locations (1):
- Universtätsklinik Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
Due to premature termination of the study, no individual participant data will be shared.